CLINICAL TRIAL: NCT01726764
Title: Is There a Pharmacokinetic Interaction Between St John's Wort and Metformin?
Brief Title: Interaction Between St John's Wort and Metformin?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Tore B. Stage, M.Sc. Pharm, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AKF-382
Record Dates: First submitted 2012-11-02; First posted 2012-11-15 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression | interventions — Hypericum extract LI 160; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): 7 days of pretreatment with metformin before full pharmacokinetics and other goals are investigated.
  Minimum 1 week of washout after this period. 3 weeks of pretreatment with St John's Wort and the last 7 days metformin is ingested again, and the same effect parameters as described above is performed again
  Interventions: Other: St John's Wort; Drug: Metformin

INTERVENTIONS:
Other: St John's Wort
Drug: Metformin

SUMMARY:
The goal of the study is to examine the difference of the pharmacokinetics of metformin with and without a 3 weeks pretreatment of St John's Wort. Furthermore secondary objectives include changes in GLP-1, C-peptide, serum-insulin and plasma-glucose during an oral glucose tolerance test, changes in OCT1 mRNA in plasma and changes in leptin and lipid-profile following this possible interaction.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-64 years
* Homozygous for common genetic variants in the genes organic cation transporter 1/2 (OCT1/OCT2)
* Normal values of biomarkers accounting for: Liver and kidney function, and normal blood glucose

Exclusion Criteria:

* Chronic alcohol abuse
* Hypersensitivity to metformin or St John's Wort
* Daily intake of drugs requiring prescription

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Area Under Curve (AUC) 0-24h of metformin | Concentration of metformin at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24 hours after metformin ingestion
  Change in 0-24h AUC of metformin after 3 weeks of treatment with St John's Wort

SECONDARY OUTCOMES:
Oral glucose tolerance test (OGTT) | During the first 2 hours of each metformin ingestion
  Changes in: Plasma-glucose, serum-insulin, glucagon-like peptide 1 (GLP-1) and connecting-peptides (C-peptides) during the oral glucose tolerance test, measured at 0, 0.5, 1, 1.5 and 2 hours after metformin ingestion.
Pharmacokinetics of metformin | Concentration of metformin at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24 hours after metformin ingestion, which will be used to determine the pharmacokinetic parameters mentioned below
  Determination of other pharmacokinetic parameters of metformin such as clearance (CL), absorption fraction (F), distribution volume (V), the minimum concentration at steady state (Css,min), elimination half life (T 1/2) etc.
Change in messenger RiboNucleic Acid (mRNA) | Will be measured 4 times: At inclusion (t=0 on that day), at t=0 in both periods and minimum 3 weeks after finalization of the study (t=0 on that day)
  Changes in mRNA encoding OCT1 will be measured at 4 different time points to give an insight to the importance of St John's Wort effect on the OCT1 production

OTHER OUTCOMES:
Hypericin/hyperforin | At t=0 in 2nd period
  If possible measure the concentrations of some of the active components of St John's Wort, hypericin and hyperforin

CONTACTS AND LOCATIONS:
Overall Officials: Per Damkier, MD ph.d., Principal Investigator — University of Southern Denmark; Tore B. Stage, M.Sc. Pharm, Principal Investigator — University of Southern Denmark; Kim Brøsen, Professor, MD, Study Director — University of Southern Denmark
Locations (1):
- Department of Clinical Pharmacology, Institute of Public Health, University of Southern Denmark, Odense, Denmark